CLINICAL TRIAL: NCT02832011
Title: The Effect on Immunological Parameters and Growth of Olive Oil and Eoprotin Used as a Fortification Breast Milk at the VLBW Babies
Brief Title: How Effect Olive Oil and Eoprotin on Immunological Parameters and Growth
Acronym: RDS
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: nihat demir (Other)
Responsible Party: Sponsor-Investigator, nihat demir, Principal Investigator, Yuzuncu Yil University
Organization: Yuzuncu Yil University (Other)
Allocation: Randomized | Model: Parallel | Masking: Single
Other Study IDs: 2015-TF-U362
Record Dates: First submitted 2016-06-29; First posted 2016-07-13 (Estimated); Last update posted 2016-07-13 (Estimated); Status verified 2016-07

CONDITIONS: Breast Milk Expression; Premature Birth of Newborn
MeSH Terms: conditions — Breast Milk Expression; Premature Birth | interventions — Olive Oil; Aptamil

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- olive oil (Active Comparator): After randomization, Investigators will give human milk fortiﬁed with olive oil
  Interventions: Dietary Supplement: olive oil; Dietary Supplement: Eoprotin
- Eoprotin (Active Comparator): After randomization, Human milk fortiﬁed with Eoprotin according to the recommendations of the manufacturer (1g per 30ml milk)
  Interventions: Dietary Supplement: olive oil; Dietary Supplement: Eoprotin

INTERVENTIONS:
Dietary Supplement: olive oil — The infants fed with olive oil will have received same amount of calorie with infants who will receive eoprotin-fortified breast milk.
  Other Names: Komili (extra virgin olive oil)
Dietary Supplement: Eoprotin — Low birth weight infants are premature infants that born with birth weight less than 1500 g. Because these infants have low birth weight, weight gain can be increased by fortifying breast milk after post-natal 7 with eoprotin.
  Other Names: aptamil

SUMMARY:
This study aims to compare immunologic parameters of 60 patients who are 1-28 days-aged, below 1500-gram body weight, born before 32 weeks of gestational age and fed with eoprotin or olive-oil fortified breast milk. Cases will receive same amount of calorie intake either with eoprotin or olive oil fortified-breast milk. If investigators identify that olive oil doesn't increase proinflammatory cytokines and grant enough weight gain in premature infants at the end of the study, investigators will suggest olive oil to replace eoprotin which is a very costly breast milk-fortifier.

DETAILED DESCRIPTION:
Low birth weight infants are premature infants that born with birth weight less than 1500 g. Because these infants have low birth weight, weight gain can be increased by fortifying breast milk after post-natal 7. day. Breast milk fortifiers might be preferred for very low birth weight or extremely low birth weight infants (infants with <1000 g birth weight infants) for faster weight gain. It does not increase risk of necrotizing enterocolitis or infection; and it has lower incidences of necrotizing enterocolitis and sepsis comparing to formula. Breast milk is usually fortified with 100 cc/kg/day enteral feeding (1,2,3,4). Even though many centers use olive oil to fortify breast milk for many years; there is no study to evaluate its scientific value. Hence it has been known that olive oil based parenteral nutrition solutions are well-tolerated by premature infants, are immunologically more neutral, does not increase proinflammatory cytokines; olive oil is the only fat consumed in its natural form and has antimicrobial and cytotoxic effects, lowers serum cholesterol concentration by decreasing cholesterol absorption, has protective measures against cardiovascular diseases due to antioxidant effects of ingredients such as mono- and poly-unsaturated fatty acids, phenolic substances, tocopherols and carotenoids; olive oil has antioxidant, cell renewal and anti- carcinogenic features because of containing squalene which is precursor of steroid synthesis and help digestion by increasing digestive juice by major pigments such as chlorophyll, pheophytin and chlorophyll (5).

In previous studies; it has been shown that nutritional support with parenteral olive oil emulsion has better plasma lipid content similarities to breast milk, lower proinflammatory cytokine synthesis, lower lipid peroxidation product levels, stronger T-cell response, higher E vitamin levels; and thus lower risk of nosocomial infections, SIRS (systemic inflammatory response syndrome), BPD (bronchopulmonary dysplasia), NEC (necrotizing enterocolitis), PVL (periventricular leukomalacia), ROP (retinopathy of prematurity) and cardiovascular diseases and positive impact on glucose metabolism. Participants hypothesize that oral olive oil intake will have similar effects (6).

Investigators aims to compare post-nutritional immunologic parameters of 1-28 day-aged 60 infants with <1500 g birth weight and < 32 weeks of gestational age who were fed with maternal milk that is fortified with eoprotin and olive oil and diagnosed and followed-up in Neonatal Intensive Care Unit of Pediatrics Department of Medicine Faculty of Yüzüncü Yıl University.

This study will be conducted on 60 patients who are 1-28 days-aged, below 1500-gram body weight, born before 32 weeks of gestational age and diagnosed and followed in Neonatal Unit of Pediatrics Department of Medicine Faculty of Yüzüncü Yıl University. For 45 days, 30 patients will receive eoprotin as breast milk fortifier while another 30 patients will receive olive oil, then 3 cc of blood will be taken from all patients at 0, 15., 30. and 45. days into biochemistry vials and will be stored at -80 C after centrifuge. At the end of the study, vials will be thawed in room temperature and serum TNF-alpha, IL-1 Beta, IL-6, IL-8, IL-10 levels will be analyzed with ELISA method by BIO-Tec ELx800 Absorbance Reader device and lipid profiles (LDL, HDL, Total cholesterol and triglyceride) and levels will be analyzed with spectrophotometric method by Architect ci16200; then these parameters will be compared with each other.

After feeding with olive oil infants will have received same amount of calorie with infants who will receive eoprotin-fortified breast milk. At the end of study, if participants identify that olive oil doesn't increase proinflammatory cytokines and provide enough weight gain in premature infants, investigators will suggest olive oil to replace eoprotin which is a very costly breast milk-fortifier. Investigators believe this situation will contribute to both country and family budgets.

ELIGIBILITY:
Inclusion Criteria:

* Infants with <1500 g birth weight
* Infants with< 32 weeks of gestational age
* Infants who will be fed with maternal milk that is fortified with eoprotin and olive oil

Exclusion Criteria:

* Critical ill patients
* Evident severe congenital malformation
* Intolerance of feeding
* Evident gastrointestinal malformation

Ages: 1 Day to 28 Days | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 60 (Estimated)
Dates: Start 2016-01; Primary Completion 2017-01 (Estimated); Study Completion 2017-06 (Estimated)

PRIMARY OUTCOMES:
serum alpha tumor necrosis factor will be analyzed | Within18 months
  For 45 days, 30 patients will receive eoprotin as breast milk fortifier while another 30 patients will receive olive oil, then 3 cc of blood will be taken from all patients at 0, 15., 30. and 45. days into biochemistry vials and will be stored at -80 C after centrifuge.
  At the end of the study, participants will be analyzed tumor necrosis factor alpha with ELISA method by BIO-Tec ELx800 Absorbance Reader device ;
IL-1 Beta will be analyzed | Within18 months
  For 45 days, 30 patients will receive eoprotin as breast milk fortifier while another 30 patients will receive olive oil, then 3 cc of blood will be taken from all patients at 0, 15., 30. and 45. days into biochemistry vials and will be stored at -80 C after centrifuge.
  At the end of the study, participants will be analyzed IL-1 with ELISA method by BIO-Tec ELx800 Absorbance Reader device ;
IL-6 will be analyzed | Within18 months
  For 45 days, 30 patients will receive eoprotin as breast milk fortifier while another 30 patients will receive olive oil, then 3 cc of blood will be taken from all patients at 0, 15., 30. and 45. days into biochemistry vials and will be stored at -80 C after centrifuge.
  At the end of the study, participants will be analyzed IL-6 with ELISA method by BIO-Tec ELx800 Absorbance Reader device ;
IL-8 will be analyzed | Within18 months
  For 45 days, 30 patients will receive eoprotin as breast milk fortifier while another 30 patients will receive olive oil, then 3 cc of blood will be taken from all patients at 0, 15., 30. and 45. days into biochemistry vials and will be stored at -80 C after centrifuge.
  At the end of the study, participants will be analyzed IL-8 with ELISA method by BIO-Tec ELx800 Absorbance Reader device ;
IL-10 will be analyzed | Within18 months
  For 45 days, 30 patients will receive eoprotin as breast milk fortifier while another 30 patients will receive olive oil, then 3 cc of blood will be taken from all patients at 0, 15., 30. and 45. days into biochemistry vials and will be stored at -80 C after centrifuge.
  At the end of the study, participants will be analyzed IL-10 with ELISA method by BIO-Tec ELx800 Absorbance Reader device ;
Triglyceride will be analyzed | Within18 months
  For 45 days, 30 patients will receive eoprotin as breast milk fortifier while another 30 patients will receive olive oil, then 3 cc of blood will be taken from all patients at 0, 15., 30. and 45. days into biochemistry vials and will be stored at -80 C after centrifuge.
  At the end of the study, participants will be analyzed triglyceride with spectrophotometric method by Architect ci16200;
Total cholesterol will be analyzed | Within18 months
  For 45 days, 30 patients will receive eoprotin as breast milk fortifier while another 30 patients will receive olive oil, then 3 cc of blood will be taken from all patients at 0, 15., 30. and 45. days into biochemistry vials and will be stored at -80 C after centrifuge.
  At the end of the study, participants will be analyzed total cholesterol with spectrophotometric method by Architect ci16200;
Low density lipoprotein (LDL) will be analyzed | Within18 months
  For 45 days, 30 patients will receive eoprotin as breast milk fortifier while another 30 patients will receive olive oil, then 3 cc of blood will be taken from all patients at 0, 15., 30. and 45. days into biochemistry vials and will be stored at -80 C after centrifuge.
  At the end of the study, participants will be analyzed Low density lipoprotein (LDL) with spectrophotometric method by Architect ci16200;
High density lipoprotein (HDL) will be analyzed | Within18 months
  For 45 days, 30 patients will receive eoprotin as breast milk fortifier while another 30 patients will receive olive oil, then 3 cc of blood will be taken from all patients at 0, 15., 30. and 45. days into biochemistry vials and will be stored at -80 C after centrifuge.
  At the end of the study, participants will be analyzed High density lipoprotein (HDL) with spectrophotometric method by Architect ci16200;

SECONDARY OUTCOMES:
SIRS (systemic inflammatory response syndrome) | Within 3 months of life
  will be defined according to National Institutes of Health criteria.
Chronic Lung Disease (CLD) | up to 36 weeks of post gestational age
  Chronic Lung Disease (CLD) will be defined according to National Institutes of Health criteria.
Patent ductus arteriosus | Within 5 days of life
  Echocardiography will be performed routinely for patent ductus arteriosus within 5 days of life
Intraventricular haemorrhage | Within 1 month of life
  We will assess for intraventricular haemorrhage higher than grade II using the Papile classification system
Necrotising enterocolitis | Within 3 months of life
  Necrotising enterocolitis with the modified Bell's classification system
Retinopathy of prematurity (ROP) | Up to 3 months of life
  Retinopathy of prematurity (ROP) defined based on the criteria of the American Academy of Pediatrics, American Academy of Ophthalmology and American Association for Pediatric Ophthalmology and Strabismus.

CONTACTS AND LOCATIONS:
Overall Officials: nihat demir, Study Director — Yuzuncu Yil University

REFERENCES:
- [Background] 1. Çelik HT, Yiğit Ş. Yenidoğan ve Prematüre Bebeklerde Parenteral Beslenmede Yenilikler. Hacettepe Tıp Dergisi 2009;40:176-189.
- [Background] 2. Gülcan H. Preterm Yenidoğanlarda Parenteral Beslenmede Yenilikler. Gaziantep Tıp Dergisi 2010;16:66-74.
- [Background] 3. Gürsoy T, Yurdakök M. Prematüre Bebeklerin Beslenmesi. Çocuk Sağlığı ve Hastalıkları Dergisi 2008;51:240-251.
- [Background] 4. Ergin H, Kılıç İ, Gürses D, Sözeri A, Özdemir C. Zenginleştirilmiş Anne Sütü (Eoprotin) Alan Prematüre Bebeklerde Vücut Ağırlığının Değişimi. ADU Tıp Fakültesi Dergisi 2000;1:9-11.
- [Result] Gawecka A, Michalkiewicz J, Kornacka MK, Luckiewicz B, Kubiszewska I. Immunologic properties differ in preterm infants fed olive oil vs soy-based lipid emulsions during parenteral nutrition. JPEN J Parenter Enteral Nutr. 2008 Jul-Aug;32(4):448-53. doi: 10.1177/0148607108319802. PMID 18596318